CLINICAL TRIAL: NCT03015805
Title: Improving Access to Substance Abuse Evidence-Based Practices for Youth in the Justice System: Strategies Used by JPOs
Brief Title: Teen Success Project
Acronym: JPO-CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: George Mason University (Other); Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Ashli Sheidow, Senior Research Scientist, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DA041434-01 (NIH)
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2025-10-21 (Actual); Status verified 2024-05

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contingency Management (Experimental): This group will receive regular probation services but will also receive the Contingency Management program for substance abuse from their juvenile probation officer during regular meetings.
  Interventions: Behavioral: Contingency Management
- Probation as Usual (Active Comparator): This group will receive regular services that are usually provided by juvenile probation officers.
  Interventions: Behavioral: Probation as Usual

INTERVENTIONS:
Behavioral: Contingency Management — Contingency Management (CM) utilizes behavior modification & cognitive behavioral strategies to target adolescent alcohol or other drug (AOD) use. Protocol components are as follows: (a) The provider introduces CM to the family and engages them in the intervention; (b) The provider conducts Antecedent-Behavior-Consequence (ABC) assessments of the youth's AOD use with the youth and caregiver; (c) Based on the results of the ABC assessments, self-management planning and drug refusal skills training are implemented by the provider in collaboration with the caregiver; (d) Concurrently, a point and level system contract is filled in by the family, which provides rewards/privileges for negative drug and alcohol tests and disincentives (e.g., extra chores) for positive tests. Until continued abstinence is achieved, components "b" through "d" are repeated; (e) The provider collaborates with the family to develop plans for sustaining long-term abstinence. Typical duration of CM is 12-16 weeks.
  Arms: Contingency Management
Behavioral: Probation as Usual — Standard services that a young person would receive while under probation supervision in the state.
  Arms: Probation as Usual

SUMMARY:
The purpose of this study is to examine the effectiveness of Juvenile Probation Officers (JPOs) delivering Contingency Management (CM) to teens on their caseload who have problems with drug use. CM has already been shown to be effective at helping teens with drug problems but CM has never been delivered by JPOs. This study will test how well it works to have JPOs deliver CM during their regular meetings with teens.

DETAILED DESCRIPTION:
Alcohol and other drug (AOD) use issues among adolescents are a major public health problem resulting in significant negative outcomes and extraordinary long-term costs. The rates of AOD use issues among youth in the justice system are twice the rates among youth without justice involvement. Further, youth with AOD issues engage in more severe delinquency and continue offending as adults, and their rate of engagement in HIV/STI sexual risk behaviors is alarming. Therefore, widespread access and delivery of effective AOD interventions to juvenile offenders is of considerable importance. Unfortunately, significant challenges exist for meeting the treatment needs of justice-involved youth. Although these youth are routinely referred to community-based providers for treatment, less than 1 in 5 are able to obtain such treatment. Further, for youth and families who are able to overcome barriers and engage with service providers, it is unlikely that they will receive an intervention that is evidence-based. In light of this context, innovative strategies clearly are needed to improve access to evidence-based practices for AOD abuse among youth in the juvenile justice system. Thus, the overriding purpose of the proposed study is to increase the access to such an evidence-based practice (Contingency Management [CM]) among youth in the juvenile justice system. This study leverages and extends the investigative team's work in CM efficacy, delivery, and technology transfer in juvenile justice settings, as well as 30+ years of collaboration with juvenile justice. We posit that juvenile probation officers (JPOs) are in an ideal position to deliver an AOD evidence-based practice to youth because of their intensive involvement and frequent contact with the youth offenders under their supervision. Further, CM is ideal for JPOs to learn and implement because it is highly specified and low in complexity relative to other AOD evidence-based practices for youth. Also, JPOs regularly monitor their probationers' substance use via frequent biological screens and implement consequences based on results, making CM consistent with JPOs' work. The proposed research randomizes JPOs to 2 conditions: CM versus control (usual JPO services), and then randomizes adolescent probationers with AOD disorders across those 2 conditions. This research would provide (1) evidence for the feasibility of JPOs to deliver an AOD abuse intervention, (2) initial evidence of clinical efficacy for JPOs as service delivery providers [to address clinical public health outcomes of AOD use, criminal activity, and HIV/STI sexual risk behaviors], and (3) identify any barriers that would need to be addressed for JPOs to deliver such services. The primary motivation for this application is the clear public health need for improving and expanding delivery of AOD interventions in the juvenile justice system. The ultimate outcome would be decreased AOD use and other public health-related behaviors (i.e., criminal behaviors, HIV/STI sexual risk behaviors) among these high-risk adolescents.

ELIGIBILITY:
There are 2 types of participants in this study: juvenile probation officers and youth.

Inclusion Criteria for juvenile probation officers:

* Employed as a juvenile probation officer within one of the participating counties
* Serving clients aged 12-18 years old with a substance abuse problem

Exclusion Criteria for juvenile probation officers:

* Not employed as a juvenile probation officer within one of the participating counties
* Not serving clients aged 12-18 years old with a substance abuse problem
* Juvenile probation officers solely assigned to a specialized caseload (e.g., sexual offense or gang unit) were excluded if they were the only one in their county with that assignment because randomization would be precluded

Inclusion Criteria for youth:

* Newly opened probation case (can have previous cases)
* 12-18 years old
* Diagnostic and Statistical Manual-5 (DSM-5) substance use disorder

Exclusion Criteria for youth:

* Pervasive intellectual or developmental disorder
* Active psychotic disorder
* Youth actively involved in a Drug Court Program at time of study recruitment

Ages Eligible for Study

* Youth: 12 Years to 18 Years
* JPOs: Any age

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 310 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline scores compared to 9 months post-Baseline Urine Drug Screens (measured at 0, 3, 6 and 9 months). | Baseline to 9 months
  The number of positive drug screens from toxicology testing for tetrahydrocannabinol (THC), synthetic THC, amphetamines, methamphetamines, opiates, phencyclidine (PCP), cocaine, benzodiazepines and alcohol metabolites (Ethyl glucuronide, Ethyl sulfate ).
Changes from Baseline scores compared to 9 months post-Baseline Substance Use and Problems (measured at 0, 3, 6 and 9 months). | Baseline to 9 months
  Frequency of substance use and substance-related problems self-reported on the Global Appraisal of Individual Needs.

SECONDARY OUTCOMES:
Changes in number and severity of criminal charges in official records in the 18 months pre-Baseline compared with 18 months post-Baseline. | 18 months pre-Baseline to 18 months post-Baseline.
  Changes from 18 months pre-Baseline in offending, measured in the number and severity of offenses in official arrest records compared to 18 months post-Baseline.
Changes from Baseline scores compared to 9 months post-Baseline Delinquent Behaviors (measured at 0, 3, 6 and 9 months). | Baseline to 9 months.
  Delinquent behaviors self-reported using the Self-Report Delinquency Scale.
Changes from Baseline scores compared to 9 months post-Baseline Sexual Risk Behaviors (measured at 0, 3, 6 and 9 months). | Baseline to 9 months.
  Sexual risk behaviors self-reported using the HIV Sexual Risk Behavior Scale.
Changes from Baseline scores compared to 9 months post-BaselineTreatment Usage (measured at 0, 3, 6 and 9 months). | Baseline to 9 months.
  The number of courses of in-patient and out-patient treatment obtained by youth for substance abuse as measured by the Structured Adolescent Interview (conducted with youth and caregiver together).
Changes from Baseline scores compared to 9 months post-Baseline Internalizing and Externalizing Behaviors (measured at 0, 3, 6 and 9 months). | Baseline to 9 months.
  The frequency of youth's internalizing and externalizing behaviors as measured using the Brief Problem Checklist (self- and parent-report).
Changes from Baseline scores compared to 31 months post-Baseline Contingency Management (CM) Adherence (measured monthly for 31 months). | Baseline to 31 months.
  Adherence to CM practices by juvenile probation officers as measured using the CM-Therapist Adherence Measure (CM-TAM) (Self-report version, Tape Coding version and Youth/Caregiver versions).
Changes from Baseline in Training Needs and Training Satisfaction scores compared to 31 months post-Baseline (measured at 0,16 and 31 months). | Baseline to 31 months.
  Scores in training needs and training satisfaction as measured by the Organizational Readiness for Change-Criminal Justice Version (completed by participating juvenile probation officers).
Changes from Baseline in attitudes towards using rewards in substance abuse treatment compared to 31 months post-Baseline (measured at 0,16 and 31 months). | Baseline to 31 months.
  Ratings on attitudes towards using rewards in substance use treatment as measured by the Provider Survey of Incentives (completed by participating juvenile probation officers).
Changes from Baseline in attitudes towards Contingency Management (CM) compared to 31 months post-Baseline (measured at 0,16 and 31 months). | Baseline to 31 months.
  Ratings on attitudes towards Contingency Management as measured by qualitative ratings of audio-taped and transcribed focus groups (focus groups involve participating juvenile probation officers).

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Cassia County Juvenile Probation, Burley, Idaho
  - Canyon County Juvenile Probation, Caldwell, Idaho
  - Gooding County Juvenile Probation, Gooding, Idaho
  - Blaine County Juvenile Probation, Hailey, Idaho
  - Jerome County Juvenile Probation, Jerome, Idaho
  - Minidoka Juvenile Probation, Rupert, Idaho
  - Lincoln County Juvenile Probation, Shoshone, Idaho
  - Twin Falls County Juvenile Probation, Twin Falls, Idaho
  - Carson City Juvenile Probation, Carson City, Nevada
  - Washoe County Juvenile Probation, Reno, Nevada
  - Deschutes County Juvenile Probation, Bend, Oregon
  - Umatilla County Juvenile Probation, Pendleton, Oregon
  - Marion County Juvenile Probation, Salem, Oregon
  - Wasco County Juvenile Probation, The Dalles, Oregon

IPD SHARING:
Plan to Share IPD: No